CLINICAL TRIAL: NCT01044394
Title: Evaluating the Effectiveness of a Same-day, Reduced Volume Polyethylene Glycol + Electrolyte Solution (PEG-ELS) Bowel Preparation for Afternoon Colonoscopies
Brief Title: Same-day, Reduced Volume Bowel Preparation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: A phase III RCT was published showing this approach is effective
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Brian Jacobson, Associate professor of medicine, Boston Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-28808
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Bowel Preparation
Keywords: colonoscopy; bowel preparation; polyethylene glycol; Quality in endoscopy; Bowel Preparation for colonoscopy
MeSH Terms: interventions — Polyethylene Glycols; Bisacodyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- same day, reduced volume PEG-ELS prep (Experimental): Patients with colonoscopies scheduled in the afternoon will complete 2 liters of PEG-ELS solution the morning of their colonoscopy.
  Interventions: Drug: polyethylene glycol (PEG-ELS) and bisacodyl tablets

INTERVENTIONS:
Drug: polyethylene glycol (PEG-ELS) and bisacodyl tablets — 2 liters of PEG-ELS and 10mg of bisacodyl tablets once the morning of the colonoscopy

SUMMARY:
We seek to evaluate whether a same day, reduced liquid volume (2liters) polyethylene glycol (PEG-ELS) bowel preparation can achieve adequate colon cleansing in patients scheduled for afternoon colonoscopies. The primary outcome will be adequacy of the bowel preparation. Secondary outcomes will include Boston Bowel Preparation Scale score, patient compliance with completing the preparation, tolerability of the preparation, willingness to repeat the preparation, side effects, duration of procedure (endoscope insertion and withdrawal times), and polyp detection.

DETAILED DESCRIPTION:
The diagnostic accuracy of colonoscopy depends on the quality of the preparation. The adequacy of the preparation determines whether complete visualization of the mucosa and identification of pathologic lesions is achieved. For reasons that are not entirely clear, colonoscopies scheduled in the afternoon have been identified as a risk factor for having an inadequate preparation. Standard bowel preparation regimens at BMC include polyethylene glycol- electrolyte solutions (PEG-ELS) in full (four liters) and reduced (two liters) forms. These laxatives are typically administered either the evening prior to the colonoscopy or in "split dose" (a portion the evening before and a portion the morning of the colonoscopy). The percent of failed colonoscopies due to a fair/poor preparation in our endoscopy unit is 17-20%. Our trial seeks to establish the efficacy and safety of a reduced volume PEG-ELS laxative given on the day of the colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* English speaking patients referred for colonoscopy.

Exclusion Criteria:

* Age < 18,
* Pregnancy,
* History of bowel resection,
* Allergy to PEG-ELS, and
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Primary outcome: adequacy of bowel preparation. | 1 year

SECONDARY OUTCOMES:
Boston Bowel Preparation Scale scores, subject compliance, subject tolerability, adverse events, colonoscopy insertion & withdrawal time, number of repeat procedures needed due to inadequate bowel preparation, polyp detection, and adenoma detection. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jacobson, MD, Principal Investigator — Boston Medicial Center Gastroenterology Department
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States